CLINICAL TRIAL: NCT06242314
Title: Comparison of The Effect of A-PRF and L-PRF Application to The Palatal Region on Quality of Life and Wound Healing After Free Gingival Graft Surgery
Brief Title: L-PRF Versus A-PRF on Palatal Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Prof.Dr. Mehmet Sağlam, Principle Investigator, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1090/2020
Record Dates: First submitted 2024-01-25; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Palate; Wound
Keywords: free gingival graft; platelet rich fibrin
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L-PRF (Experimental): L-PRF was laid directly on the palatal wound immediately after free gingival graft harvesting and stabilized with silk suture.
  Interventions: Procedure: L_PRF
- A-PRF (Experimental): A-PRF was laid directly on the palatal wound immediately after free gingival graft harvesting and stabilized with silk suture.
  Interventions: Procedure: A-PRF
- Palatal stent (Placebo Comparator): Palatal stent was prepared by taking impression of the palate before surgery. After FGG harvesting, periodontal paste (COE-PAK periodontal dressing, GC, Illinois, USA) was applied on the wound surface of the palatal stent and the palate was closed.
  Interventions: Procedure: Palatal stent

INTERVENTIONS:
Procedure: L_PRF — Palatal epithelialization, pain (Visual Analog Scale (VAS) recording), analgesic tablet use and Oral Health Impact Proﬁle-14 (OHIP-14) questionnaire scores were recorded after L-PRF placing on palatal wounds
  Arms: L-PRF
Procedure: A-PRF — Palatal epithelialization, pain (Visual Analog Scale (VAS) recording), analgesic tablet use and Oral Health Impact Proﬁle-14 (OHIP-14) questionnaire scores were recorded after A-PRF placing on palatal wounds
  Arms: A-PRF
Procedure: Palatal stent — Palatal epithelialization, pain (Visual Analog Scale (VAS) recording), analgesic tablet use and Oral Health Impact Proﬁle-14 (OHIP-14) questionnaire scores were recorded after palatal stent placing on palatal wounds
  Arms: Palatal stent

SUMMARY:
Different approaches are used to reduce post-operative complications associated with the palatal wound site after free gingival graft (FGG) harvesting. The aim of this study was to compare the effects of L-PRF and A-PRF on palatal wound healing after free gingival graft harvesting and patients' quality of life.

DETAILED DESCRIPTION:
Thirty-six patients between the ages of 18 and 60 years (11 males and 25 females) who had completed Phase 1 periodontal treatments and for whom FGG surgery was indicated for isolated gingival recession defects limited to one or two teeth with shallow vestibule and insufficient keratinized or attached gingival width were included in the present study.

Three different treatments were performed on palatal wound areas: L-PRF (L-PRF group, n = 12), A-PRF (A-PRF group, n = 12) and palatal stent (control group, n = 12) OHIP-14 scores, VAS scores (for pain), analgesic tablet intake, and epithelialization condition were recorded for different time points.

ELIGIBILITY:
Inclusion Criteria:

• Patients ≥18 years requiring FGG surgery because of shallow vestibule and insufficient keratinized/attached gingival width

Exclusion Criteria:

* no smoking /no alcohol use,
* not suffering from any systemic disease that could impair the healing of wounds,
* pregnancy or lactation,
* Previous graft harvesting from the same site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Epithelialization | 1 month
  Hydrogen peroxide (H2O2) test was used to evaluate the integrity of epithelialization

SECONDARY OUTCOMES:
Pain at Palatal wound area | First 7 days and day 14
  Postoperative pain was evaluated using a 10-cm Visual Analog Scale (VAS) score during the first week and on day 14. The left end-point represented "no pain," while the right end-point represented "severe pain at its highest." In order to rate their pain, the participants were requested to indicate the VAS line with the appropriate postoperative pain level. A ruler was then used to measure the distance between the "no pain" point and the rated line, providing a pain score between 0 and 10
Pain at Palatal wound area | First 7 days
  The average amount of ibuprofen 600 mg pills needed to control postoperative discomfort during the seven days after surgery was recorded as the total number of pills consumed.
Oral health-related quality of life (OHRQoL) | 7 and 14 days after free gingival graft surgery
  Oral health-related quality of life of patients was assessed by the Oral Health Impact Proﬁle-14 (OHIP-14) questionnaire.OHIP-14 uses 14 structured questions and answers to assess seven subjective dimensions. The evaluated dimensions are functional limitations, physical pain, psychologic discomfort, physical disability, psychologic disability, social disability, and handicap. Patients responded to the questionnaire using Likert scale answers (0- never; 1-almost never; 2-occasionally; 3-quite frequent; 4-very common) on the 7th and 14th day after surgery. In this way, the questionnaire ranges from 0 to 56 points, with higher scores indicating more negative impact of oral conditions on quality of life.Thus, patients' experiences about the surgery in the first two weeks postoperatively were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Sağlam, Izmir, Çiğli, Turkey (Türkiye)